CLINICAL TRIAL: NCT06878144
Title: MD Anderson Mucormycosis Clinical Core for the MUCOR-ADVANCE P01 Project (Deciphering Immunopathogenesis of MUCORmycosis to ADVANCE Risk Stratification, Diagnosis and Management of the Disease)
Brief Title: Mucormycosis Clinical Core for the MUCOR-ADVANCE P01 Project
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-1965; NCI-2025-01921 (Other: NCI -CTRP Clinical Registry)
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Mucormycosis
MeSH Terms: conditions — Mucormycosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Group M: Patients with mucormycosis undergo collection of blood, tissue and BAL fluid samples as well as have their medical records reviewed on study.
  Interventions: Behavioral: Mucormycosis
- Group A: Patients with mucormycosis undergo collection of blood, tissue and BAL fluid samples as well as have their medical records reviewed on study.
  Interventions: Behavioral: Mucormycosis
- Group B: Patients with mucormycosis undergo collection of blood, tissue and BAL fluid samples as well as have their medical records reviewed on study.
  Interventions: Behavioral: Mucormycosis
- Group C: Patients with mucormycosis undergo collection of blood, tissue and BAL fluid samples as well as have their medical records reviewed on study.
  Interventions: Behavioral: Mucormycosis

INTERVENTIONS:
Behavioral: Mucormycosis — Tell the study team about any symptoms or side effects you have, follow study directions, and come to all study appointments (or contact the study team to reschedule).

SUMMARY:
To collect data and samples from participants with cancer who also have invasive mucormycosis, invasive aspergillosis, bacterial pneumonia, or a risk for fungal infection.

DETAILED DESCRIPTION:
Primary Objective:

To establish MD Anderson Mucormycosis Clinical Core for the MUCOR-ADVANCE P01 Project.

* To prospectively identify, collect, and store all isolates causing proven or probable MCM in adult high-risk cancer participants.
* To prospectively identify, collect, and store relevant host samples from high-risk participants developing proven or probable MCM, along with relevant biospecimens from three control groups.
* To comprehensively annotate clinical specimens and provide information regarding the course and outcome of all MCM cases and controls.

OUTLINE:

This is an observational study. Patients are assigned to 1 of 4 groups.

GROUP M: Patients with mucormycosis undergo collection of blood, tissue and BAL fluid samples as well as have their medical records reviewed on study.

GROUP A: Patients with mucormycosis undergo collection of blood, tissue and BAL fluid samples as well as have their medical records reviewed on study.

GROUP B: Patients with mucormycosis undergo collection of blood, tissue and BAL fluid samples as well as have their medical records reviewed on study.

GROUP C: Patients with mucormycosis undergo collection of blood, tissue and BAL fluid samples as well as have their medical records reviewed on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18-100 years old and have cancer and invasive mucormycosis, invasive aspergillosis, bacterial pneumonia, or a risk for fungal infection but no evidence of such infection.
* Patients must be willing to undergo routine diagnostic procedures (e.g., phlebotomy, bronchoscopy, biopsy) as part of their regular care.

Exclusion Criteria:

• Patients who are unwilling to undergo routine diagnostic procedures as part of their regular care.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-30 (Estimated); Primary Completion 2030-12-31 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Kontoyiannis, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org